CLINICAL TRIAL: NCT02309086
Title: Phase I-II Vaccination Clinical Trial in Patients With Chronic Hepatitis C by Administration of Autologous Dendritic Cells Transduced With an Adenoviral Vector Encoding NS3 Protein
Brief Title: Phase I-II Vaccination of Autologous Dendritic Cells Transduced With Adenoviral Vector Encoding NS3 in Hepatitis C Encoding NS3 in Hepatitis C
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Centro de Investigación Médica Aplicada (CIMA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-AdNS3
Record Dates: First submitted 2014-11-18; First posted 2014-12-05 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Autologous dendritic cells transduced with Ad encoding NS3
  Interventions: Biological: Autologous dendritic cells transduced with Ad encoding NS3

INTERVENTIONS:
Biological: Autologous dendritic cells transduced with Ad encoding NS3 — Patients will receive 3 different dosis of the vaccine via subcutaneous injection

SUMMARY:
Dendritic cells (DC) play a central role in the activation of T-cell responses and have shown to be very immunogenic in preclinical in vivo and in vitro assays. The aims of this study is to assess the efficacy of therapeutic vaccination pilot clinical trial in Genotype 1 HCV patients using autologous DC transduced with a recombinant adenovirus encoding NS3

ELIGIBILITY:
Inclusion Criteria:

Chronic hepatitis C (genotype 1b) that had previously failed Interferon/Ribavirin-based treatment

Exclusion Criteria:

Liver cirrhosis HBV-coinfection Bilirubin >1.5 times ULN or ALT >7 ULN Hepatocellular carcinoma Immunodeficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability determined by the evaluation of the number of participants with the type adverse events. Liver safety will be assessed by blood analysis and Ultrasound. | 6 months
  Safety assessment will be determined by the evaluation of the number of participants with the type adverse events. Liver safety will be assessed by blood analysis and Ultrasound.

SECONDARY OUTCOMES:
Efficacy on viral load and immune response | 6 months